CLINICAL TRIAL: NCT03947411
Title: A Multicenter, Randomized, Open Label, Add-on Study to Assess Efficacy and Safety of Xiyanping Injection in Pediatric Participants With Severe Influenza-Like Symptoms
Brief Title: Evaluate the Safety and Efficacy of Xiyanping in Pediatric Participants With Severe Influenza-Like Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); Beijing Luhe Hospital (Other); Qingdao Municipal Hospital (Other); Cangzhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JXQF- XYP-1801
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Severe Influenza
Keywords: severe Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oseltamivir Phosphate+Xiyanping injection (Experimental): Oseltamivir Phosphate+Xiyanping injection treatment for 7-10 days
  Interventions: Drug: Xiyanping injection+Oseltamivir Phosphate
- Oseltamivir Phosphate treatment only (Active Comparator): Oseltamivir Phosphate treatment for 7-10 days
  Interventions: Drug: Oseltamivir Phosphate

INTERVENTIONS:
Drug: Oseltamivir Phosphate — Take the dosage of Oseltamivir Phosphate recommended according to the instructions.support treatment such as antiasthmatic, expectorant and antipyretic use only in need.
  Arms: Oseltamivir Phosphate treatment only
Drug: Xiyanping injection+Oseltamivir Phosphate — Take the dosage of Oseltamivir Phosphate recommended according to the instructions.Xiyanping injection intravenous administration of 0.4mL/kg/day ,QD for 7-10 days.support treatment such as antiasthmatic, expectorant and antipyretic use only in need.
  Arms: Oseltamivir Phosphate+Xiyanping injection

SUMMARY:
This is a multicenter, randomized, open Label, add-on study.

DETAILED DESCRIPTION:
This is an add-on study of efficacy and safety of intravenous injection of Xiyanping injection in pediatric subjects with severe Influenza-Like Symptoms.

The purpose to determine the efficacy and safety of Oseltamivir Phosphate combined with or without Xiyanping injection in the treatment of severe Influenza-Like Symptoms. The study will enroll 72 Pediatric severe Influenza-Like Symptoms volunteers, who will be randomized into 2 groups (1:1 ratio): volunteers from the first group will receive Oseltamivir Phosphate and Xiyanping injection for severe Influenza; volunteers from the second group will receive Oseltamivir Phosphate for severe Influenza. Xiyanping injection will be administration as intravenous injection of 0.4mL/kg/day once daily for 7-10 days concomitantly with Oseltamivir Phosphate for severe Influenza-Like Symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 6 years old;
* Clinical diagnosis of Severe Influenza with hospital treatment needed;
* Patients did not accept oseltamivir phosphate treatment or symptoms persisted for more than 3 days treatment;

  （1)Fever ≥ 39°C (tympanic temperature) for at least 3 days with Severe cough,sputum, blood stasis, or chest pain; （2）Combined pneumonia;
* The rapid viral antigen test of throat swab and nose swab results were positive;
* Guardians understood and assigned the informed consent;

Exclusion Criteria:

* Participants allergenic to XiYanPing injection, Andrographolide or Oseltamivir Phosphate;
* Creatinine clearance <80ml/min or received continuous renal replacement therapy (CRRT) test;
* Need extracorporeal membrane oxygenation (ECMO) at baseline;
* Glasgow Coma Rating Scale (GCS) score ≤ 9 points when dyspnea, altered consciousness, severe vomiting, or coma appeared at baseline;
* Crisis influenza Symptoms, such as respiratory failure, acute necrotizing encephalopathy, septic shock, multiple organ dysfunction and other serious clinical conditions requiring monitoring;
* Use of systemic steroids or other immunosuppressants;
* Participants with the following underlying diseases, including: heart disease (such as New York Heart Function Classification II-IV) or clinically significant arrhythmia (such as QTc ≥ 480ms), malignant tumor or other malignant diseases, autoimmune diseases; liver and kidney diseases ( ALT and AST ≥ 1.5 × ULN; Cr and BUN > 1.2 × ULN), blood diseases, nervous system diseases, immune system diseases and endocrine diseases, consciousness, speech, behavioral abnormalities caused by encephalitis / encephalopathy or limb paralysis, severe malnutrition, etc.
* Participants used Influenza virus vaccine within 3 months;
* Participants with drug dependence or with mental disorders within 1 year;
* Participants participated in other clinical research in the last 30 days;
* Any condition which would make the subject, in the opinion of the investigator or designee, not suitable for the study for any reason.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — 3 to 6 years old hospitalized patient
Enrollment: 72 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to Alleviation of Influenza Signs and Symptoms | Up to Day 12
  Time to alleviation of influenza signs and symptoms is defined as the length of time taken from the start of treatment to the point at which all of the signs and symptoms are alleviation or recovery.
Duration of Fever | Up to Day 12
  Length of time taken by participants to return to afebrile state

SECONDARY OUTCOMES:
Signs and Symptoms Score from baseline | Up to Day 12
  (1) recovery: symptom score reduction rate ≥ 95%; (2) markedly effective: symptom score reduction rate ≥ 70%; (3) progress: symptom score reduction rate ≥ 30%; (4) invalid: Symptom score reduction rate <30%.
Usage of antibiotic,hormone and incidence of critical cases | Up to Day 12
Time to Cessation of Viral Shedding by RT-PCR | Up to Day 12
Relief time of individual symptom such as:expectoration, cough | Up to Day 12
Disease efficacy criteria | Up to Day 12
  (1) Healing: The body temperature is normal within 48 hours of treatment, the symptoms disappeared without repetition. (2) markedly effective: the body temperature is normal within 48 hours of treatment, and the symptom score is reduced by more than 2/3. (3) Effective: The body temperature is normal within 72 hours of treatment, and the remaining symptom scores are reduced by 2/3-1/3. (4) Invalid: The condition did not improve or worsened after 72 hours of treatment.
Imaging improvement rate: number of people with normal or baseline imaging | Up to Day 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided